CLINICAL TRIAL: NCT01009086
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Ustekinumab, a Fully Human Aanti-IL-12/23p40 Monoclonal Antibody, Administered Subcutaneously, in Subjects With Active Psoriatic Arthritis
Brief Title: A Study of the Safety and Effectiveness of Ustekinumab in Patients With Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016315; CNTO1275PSA3001 (Other: Janssen Research & Development, LLC); 2009-012264-14 (EudraCT Number); NCT01902706 (obsolete NCT alias)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Arthritis, Psoriatic
Keywords: Arthritis, Psoriatic; Ustekinumab; CNTO 1275; Stelara; Psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Experimental): Participants will receive subcutaneous (SC) injections of placebo at Weeks 0, 4, 16, and 20. At Week 24 participants will cross over to receive SC injections of ustekinumab 45 mg at Weeks 24 and 28 and every 12 weeks thereafter with the last dose at Week 88. If early escape, SC injections of 45 mg ustekinumab will be given at Weeks 16, 20, and 28 and every 12 weeks thereafter with the last dose at Week 88. For participants entering early escape, a SC placebo injection will be given at Week 24 to maintain the blind.
  Interventions: Drug: Placebo
- Ustekinumab 45 mg (Experimental): Participants will receive SC injections of ustekinumab 45 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 88. If early escape, SC injections of 90 mg ustekinumab will be given at Week 16 and every 12 weeks thereafter with the last dose at Week 88. Participants will receive SC injections of placebo at Weeks 20 and 24 to maintain the blind.
  Interventions: Drug: Placebo; Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg
- Ustekinumab 90 mg (Experimental): Participants will receive SC injections of ustekinumab 90 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 88. If early escape, the same dosage schedule will continue. Participants will receive SC injections of placebo at Weeks 20 and 24 to maintain the blind.
  Interventions: Drug: Placebo; Drug: Ustekinumab 90 mg

INTERVENTIONS:
Drug: Placebo — SC injections
Drug: Ustekinumab 45 mg — SC injections
  Arms: Ustekinumab 45 mg
Drug: Ustekinumab 90 mg — SC injections
  Arms: Ustekinumab 45 mg; Ustekinumab 90 mg

SUMMARY:
The purpose of this study is to evaluate the effectiveness (improvement of signs and symptoms) and safety of ustekinumab in participants with active psoriatic arthritis.

DETAILED DESCRIPTION:
This is a randomized (participants are assigned different treatments based on chance), double-blind (neither the participant nor the physician knows whether drug or placebo is being taken, or at what dosage), parallel-group (each group of participants will be treated at the same time), and multicenter (study conducted at multiple sites) study. Approximately, 615 participants will participate in this study. Participants will be assigned to one of three treatment groups: Group I: ustekinumab 45 mg, Group II: ustekinumab 90 mg, and Group III: placebo group (an inactive substance). Participants will receive either 45 mg ustekinumab or 90 mg ustekinumab at Weeks 0, 4, and every 12 weeks until Week 88 as randomized to respective groups. Participants in placebo group will receive placebo at Weeks 0, 4, 16, and 20 and 45 mg ustekinumab at Weeks 24 and 28 followed by every 12 weeks dosing until Week 88. Participants who do not have greater than or equal to 5 percentage improvement in their disease (tender and swollen joints) will be eligible for an early escape. Specifically, during early escape at Week 16, participants in Group I will receive 90 mg ustekinumab, for participants in Group II same dosing schedule will be continued, and participants in placebo group will receive 45 mg ustekinumab. Safety evaluations will include assessments of adverse events, clinical laboratory tests, and physical examination. The maximum study duration will be approximately 108 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have had a documented diagnosis of psoriatic arthritis (PsA) at least 6 months
* Have a diagnosis of active PsA at the time of entry into the study
* If the participant is using methotrexate they should have started treatment at a dose not to exceed 25 milligram per week at least 3 months prior to the beginning of the study and should have no serious toxic side effects attributable to methotrexate. Methotrexate route of administration and doses should be stable for at least 4 weeks prior to the first administration of study agent. If currently not using methotrexate, must have not received methotrexate for at least 4 weeks prior to the first administration of the study agent

Exclusion Criteria:

* Have other inflammatory diseases, including but not limited to rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, or Lyme disease
* Have used any therapeutic agent targeted at reducing interleukin (IL)-12 or IL-23, including but not limited to ustekinumab and briakinumab (ABT-874)
* Have used any biologic agents that are targeted for reducing tumor necrosis factor-alpha, including but not limited to infliximab, etanercept, adalimumab, and golimumab
* Have a medical history of latent or active granulomatous infection
* Have any known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years of the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (102):
- United States (26):
  - Encinitas, California
  - La Jolla, California
  - San Diego, California
  - Denver, Colorado
  - Trumbull, Connecticut
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Worcester, Massachusetts
  - Edina, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Freehold, New Jersey
  - Norman, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Jackson, Tennessee
  - Houston, Texas
  - Webster, Texas
  - Seattle, Washington
- Australia (6):
  - Camperdown
  - Heidelberg
  - Maroochydore
  - Melbourne
  - Perth
  - Woodville
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Canada (18):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - North Bay, Ontario
  - Saint Catherines, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Québec, Quebec
  - Trois-Rivières, Quebec
  - Westmount, Quebec
- Finland (2):
  - Helsinki
  - Hyvinkää
- Germany (9):
  - Berlin
  - Frankfurt
  - Hamburg
  - Herne
  - Kiel
  - Mahlow
  - Mainz
  - Regensburg
  - Tübingen
- Hungary (6):
  - Budapest
  - Debrecen
  - Kecskemét
  - Szeged
  - Szolnok
  - Veszprém
- Riga, Latvia
- Lithuania (4):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
- New Zealand (4):
  - Auckland
  - Christchurch
  - Rotorua
  - Wellington
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Lublin
  - Torun
  - Warsaw
- Russia (7):
  - Korolyov
  - Moscow
  - Novosibirsk
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Yekaterinburg
- Spain (4):
  - Barcelona
  - Oviedo
  - Santiago de Compostela
  - Seville
- United Kingdom (6):
  - Cannock
  - Glasgow
  - London
  - Metropolitan Borough of Wirral
  - Salford
  - Wigan

REFERENCES:
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Ustekinumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1413-1423. doi: 10.1007/s40744-024-00705-x. Epub 2024 Aug 9. PMID 39120848
- [Derived] Helliwell PS, Gladman DD, Chakravarty SD, Kafka S, Karyekar CS, You Y, Campbell K, Sweet K, Kavanaugh A, Gensler LS. Effects of ustekinumab on spondylitis-associated endpoints in TNFi-naive active psoriatic arthritis patients with physician-reported spondylitis: pooled results from two phase 3, randomised, controlled trials. RMD Open. 2020 Feb;6(1):e001149. doi: 10.1136/rmdopen-2019-001149. PMID 32209721
- [Derived] Siebert S, Sweet K, Dasgupta B, Campbell K, McInnes IB, Loza MJ. Responsiveness of Serum C-Reactive Protein, Interleukin-17A, and Interleukin-17F Levels to Ustekinumab in Psoriatic Arthritis: Lessons From Two Phase III, Multicenter, Double-Blind, Placebo-Controlled Trials. Arthritis Rheumatol. 2019 Oct;71(10):1660-1669. doi: 10.1002/art.40921. Epub 2019 Sep 3. PMID 31070869
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Rahman P, Puig L, Gottlieb AB, Kavanaugh A, McInnes IB, Ritchlin C, Li S, Wang Y, Song M, Mendelsohn A, Han C; PSUMMIT 1 and 2 Study Groups. Ustekinumab Treatment and Improvement of Physical Function and Health-Related Quality of Life in Patients With Psoriatic Arthritis. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1812-1822. doi: 10.1002/acr.23000. Epub 2016 Oct 21. PMID 27483458
- [Derived] Kavanaugh A, Puig L, Gottlieb AB, Ritchlin C, You Y, Li S, Song M, Randazzo B, Rahman P, McInnes IB. Efficacy and safety of ustekinumab in psoriatic arthritis patients with peripheral arthritis and physician-reported spondylitis: post-hoc analyses from two phase III, multicentre, double-blind, placebo-controlled studies (PSUMMIT-1/PSUMMIT-2). Ann Rheum Dis. 2016 Nov;75(11):1984-1988. doi: 10.1136/annrheumdis-2015-209068. Epub 2016 Apr 20. PMID 27098404
- [Derived] Kavanaugh A, Puig L, Gottlieb AB, Ritchlin C, Li S, Wang Y, Mendelsohn AM, Song M, Zhu Y, Rahman P, McInnes IB; PSUMMIT 1 Study Group. Maintenance of Clinical Efficacy and Radiographic Benefit Through Two Years of Ustekinumab Therapy in Patients With Active Psoriatic Arthritis: Results From a Randomized, Placebo-Controlled Phase III Trial. Arthritis Care Res (Hoboken). 2015 Dec;67(12):1739-49. doi: 10.1002/acr.22645. PMID 26097039
- [Derived] McInnes IB, Kavanaugh A, Gottlieb AB, Puig L, Rahman P, Ritchlin C, Brodmerkel C, Li S, Wang Y, Mendelsohn AM, Doyle MK; PSUMMIT 1 Study Group. Efficacy and safety of ustekinumab in patients with active psoriatic arthritis: 1 year results of the phase 3, multicentre, double-blind, placebo-controlled PSUMMIT 1 trial. Lancet. 2013 Aug 31;382(9894):780-9. doi: 10.1016/S0140-6736(13)60594-2. Epub 2013 Jun 13. PMID 23769296

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: PLACEBO: Placebo Subcutaneous (SC) injections at Weeks 0, 4, 16 and 20. If Early Escape then participants would receive Ustekinumab 45 mg injections starting Week 16 with the last dose at Week 88. If Crossover then participants would receive Ustekinumab 45 milligram (mg) injections starting Week 24 with the last dose at Week 88.
- Group 2: USTEKINUMAB 45 MG: Ustekinumab Subcutaneous (SC) injections of 45 mg starting at Week 0 with the last dose at Week 88. If Early Escape then participants would receive Ustekinumab 90 mg injections starting Week 16 with the last dose at Week 88.
- Group 3: USTEKINUMAB 90 MG: Ustekinumab Subcutaneous (SC) injections of 90 mg starting at Week 0 with the last dose at Week 88.
Period: Overall Study
Arm/Group | Group 1: PLACEBO | Group 2: USTEKINUMAB 45 MG | Group 3: USTEKINUMAB 90 MG
Started | 206 | 205 | 204
Completed | 162 | 158 | 170
Not Completed | 44 | 47 | 34
Not completed — Lack of Efficacy | 16 | 15 | 9
Not completed — Lost to Follow-up | 4 | 5 | 3
Not completed — Adverse Event | 12 | 11 | 8
Not completed — Withdrawal by Subject | 9 | 11 | 13
Not completed — Other | 3 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: PLACEBO | Group 2: USTEKINUMAB 45 MG | Group 3: USTEKINUMAB 90 MG | Total
Number analyzed (Participants) | 206 | 205 | 204 | 615
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.29) | 47.1 (12.64) | 46.8 (11.75) | 47.1 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 99 | 88 | 285
  Male | 108 | 106 | 116 | 330

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 24.
Description: An ACR 20 response is defined as a greater than or equal to 20 percent improvement from baseline in swollen (66 joints) and tender (68 joints) joint counts and greater than or equal to 20 percent improvement in 3 of the following 5 assessments: 1) Participant's assessment of pain by Visual Analog Scale (VAS) (0-10 cm), 2) Participant's global assessment of disease activity by VAS (0-10 cm), 3) Physician's global assessment of disease activity by VAS (0-10 centimeters [cm]) 4) Participant's assessment of physical function as measured by the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI) (score of 0-3 in 8 functional areas) and 5) C reactive protein.
Time Frame: Week 24
Population: All participants randomly assigned to a treatment group were included in the efficacy analysis regardless of whether they received the assigned treatment. For early escape, data at or prior to Week 16 were carried forward through Week 24.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Participants received subcutaneous injections of placebo at Weeks 0, 4, 16, and 20. At Week 24 participants crossed over to receive subcutaneous injections of ustekinumab 45 milligram (mg) at Weeks 24 and 28 and every 12 weeks thereafter with the last dose at Week 88. If early escape, subcutaneous injections of 45 mg ustekinumab were given at Weeks 16, 20, and 28 and every 12 weeks thereafter with the last dose at Week 88. For participants entering early escape, a subcutaneous placebo injection was given at Week 24 to maintain the blind.
- Ustekinumab 45 mg: Participants received subcutaneous injections of ustekinumab 45 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 88. If early escape, subcutaneous injections of 90 mg ustekinumab were given at Week 16 and every 12 weeks thereafter with the last dose at Week 88. Participants received subcutaneous injections of placebo at Weeks 20 and 24 to maintain the blind.
- Ustekinumab 90 mg: Participants received subcutaneous injections of ustekinumab 90 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 88. Participants received subcutaneous injections of placebo at Weeks 20 and 24 to maintain the blind.
- All Ustekinumab Combined: Participants who received subcutaneous injections of ustekinumab at any dose (45 mg and 90 mg) through Week 88.
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 206 | 205 | 204 | 409
Percentage of participants | 22.8 | 42.4 | 49.5 | 46.0
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

2. Secondary Outcome: Change From Baseline to Week 24 in the Disability Index Score as Measured With the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI)
Description: The HAQ-DI is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty), to 3 (inability to perform a task in that area). The average score across the functional areas yields an overall HAQ-DI score which ranges from 0 (no disability) to 3 (completely disabled). In psoriatic arthritis, a decrease in score of 0.30 indicates clinically meaningful improvement.
Time Frame: Day 1 (Baseline) and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 206 | 205 | 204 | 409
Score on a scale | -0.10 (0.390) | -0.31 (0.521) | -0.40 (0.514) | -0.36 (0.518)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

3. Secondary Outcome: Percentage of Participants (With >= 3% Baseline Body Surface Area (BSA) Psoriatic Involvement) Who Achieved a Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 24
Description: The PASI is a physician-administered assessment tool used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). A PASI 75 response is defined as greater than or equal to 75 percent improvement in PASI score from baseline.
Time Frame: Week 24
Population: All participants randomly assigned to a treatment group, regardless of whether they received the assigned treatment. For early escape, data at or prior to Week 16 were carried forward through Week 24. Only participants with >=3% baseline BSA psoriatic involvement were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 146 | 145 | 149 | 294
Percentage of participants | 11.0 | 57.2 | 62.4 | 59.9
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50 Response at Week 24
Description: An ACR 50 response is defined as a greater than or equal to 50 percent improvement from baseline in swollen (66 joints) and tender (68 joints) joint counts and greater than or equal to 50 percent improvement in 3 of the following 5 assessments: 1) Participant's assessment of pain by Visual Analog Scale (VAS) (0-10 cm), 2) Participant's global assessment of disease activity by VAS (0-10 cm), 3) Physician's global assessment of disease activity by VAS (0-10 cm) 4)Participant's assessment of physical function as measured by the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI) (score of 0-3 in 8 functional areas) and 5) C reactive protein.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 206 | 205 | 204 | 409
Percentage of participants | 8.7 | 24.9 | 27.9 | 26.4
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

5. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70 Response at Week 24
Description: An ACR 70 response is defined as a greater than or equal to 70 percent improvement from baseline in swollen (66 joints) and tender (68 joints) joint counts and greater than or equal to 70 percent improvement in 3 of the following 5 assessments: 1) Participant's assessment of pain by Visual Analog Scale (VAS) (0-10 cm), 2) Participant's global assessment of disease activity by VAS (0-10 cm), 3) Physician's global assessment of disease activity by VAS (0-10 cm) 4) Participant's assessment of physical function as measured by the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI) (score of 0-3 in 8 functional areas) and 5) C reactive protein.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 206 | 205 | 204 | 409
Percentage of participants | 2.4 | 12.2 | 14.2 | 13.2
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

6. Secondary Outcome: Change From Baseline to Week 24 in Total Modified Van Der Heijde-Sharp (vdH-S) Score for the Combined Radiographic Data From Studies CNTO1275PSA3001 and CNTO1275PSA3002
Description: The modified vdH-S score is a radiographic evaluation of hand and feet erosions and joint space narrowing (JSN) for 20 joints per hand and 6 joints per foot with a total score ranging from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score and positive score changes indicate more radiographic damage and radiographic progression, respectively. As per protocol, analysis for this outcome measure used pooled data from 2 studies (CNTO1275PSA3001 and PSA3002) because initial power assumptions showed that 900 participants would be required to evaluate impact of ustekinumab on structural damage (SD) progression. The 2 studies, (which had similar study designs and dosing regimens with difference to prior exposure to anti-tumor necrosis factor alpha (TNFα) therapies), were intended to independently measure efficacy in terms of signs, symptoms and physical function, while effects on SD progression is provided from an integrated analysis.
Time Frame: Day 1 (Baseline) and Week 24
Population: Analysis included: (1) combined data from studies CNTO1275PSA3001 (NCT01009086) and CNTO1275PSA3002 (NCT01077362) and (2) all participants randomly assigned to a treatment group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 310 | 308 | 309 | 617
Score on a scale | 0.97 (3.852) | 0.40 (2.110) | 0.39 (2.403) | 0.40 (2.260)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p = 0.017, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

ADVERSE EVENTS:
Time Frame: Baseline up to Week 108
Description: Safety population included all participants who received the investigational drug and had safety data.
Groups:
- Placebo (CP): Controlled period (Week 0-16) - Placebo group. Placebo Subcutaneous (SC) injections will be received at Weeks 0, 4 and 16.
- Ustekinumab 45 mg (CP): Controlled period (Week 0-16) - Ustekinumab 45 mg group. Participants received SC injections of ustekinumab 45 mg at Weeks 0 and 4 and 16.
- Ustekinumab 90 mg (CP): Controlled period (Week 0-16) - Ustekinumab 90 mg group. Participants received SC injections of ustekinumab 90 mg at Weeks 0 and 4 and 16.
- Placebo (After CP): After Controlled period (Week 16-24) - participants receiving placebo at Weeks 0, 4, 16, and 20, then crossed over to ustekinumab 45 mg at Week 24.
- Placebo -> Ustekinumab 45 mg (After CP): After Controlled period (Week 16-108) - participants randomized to placebo who early escaped to ustekinumab 45 mg at Week 16 or who crossed over to ustekinumab 45 mg at Week 24.
- Ustekinumab 45 mg (After CP): After Controlled period (Week 16-108) - participants randomized to ustekinumab 45 mg at Week 0, irrespective of their early escape status.
- Ustekinumab 90 mg (After CP): After Controlled period (Week 16-108) - participants randomized to ustekinumab 90 mg at Week 0, irrespective of their early escape status.
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo (After CP) | Placebo -> Ustekinumab 45 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 4/205 | 5/205 | 3/204 | 2/140 | 14/189 | 20/203 | 13/199
Other Adverse Events (participants affected / at risk) | 30/205 | 17/205 | 29/204 | 7/140 | 50/189 | 42/203 | 57/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=205) | Ustekinumab 45 mg (CP) (N=205) | Ustekinumab 90 mg (CP) (N=204) | Placebo (After CP) (N=140) | Placebo -> Ustekinumab 45 mg (After CP) (N=189) | Ustekinumab 45 mg (After CP) (N=203) | Ustekinumab 90 mg (After CP) (N=199)
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia Mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Finger Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervical Polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=205) | Ustekinumab 45 mg (CP) (N=205) | Ustekinumab 90 mg (CP) (N=204) | Placebo (After CP) (N=140) | Placebo -> Ustekinumab 45 mg (After CP) (N=189) | Ustekinumab 45 mg (After CP) (N=203) | Ustekinumab 90 mg (After CP) (N=199)
Nasopharyngitis (Infections and infestations) | 8 | 8 | 11 | 2 | 15 | 18 | 20
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 5 | 9 | 2 | 16 | 14 | 12
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 2 | 1 | 6 | 4 | 11
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 7 | 0 | 4 | 0 | 10 | 6 | 9
Hypertension (Vascular disorders) | 4 | 3 | 6 | 2 | 7 | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.